CLINICAL TRIAL: NCT05868538
Title: Evaluation of Calprotectin and Ischemia Modified Albumin Serum Levels as Biomarkers to Measure Disease Activity in Behçet's Disease
Brief Title: Calprotectin and Ischemia Modified Albumin Serum to Measure Disease Activity in Behçet's Disease
Status: Completed | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: R.22.10.1905 - 2022/10/17
Record Dates: First submitted 2023-05-04; First posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Behçet's Diseasecases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients
  Interventions: Diagnostic Test: Serum calprotectin and IMA concentrations
- control
  Interventions: Diagnostic Test: Serum calprotectin and IMA concentrations

INTERVENTIONS:
Diagnostic Test: Serum calprotectin and IMA concentrations — Serum calprotectin and IMA concentrations were compared among active BD cases, inactive BD cases and control subjects.

SUMMARY:
Behçet's Disease activity was evaluated using BD Current Activity Form (BDCAF). Serum calprotectin and IMA concentrations were compared among active BD cases, inactive BD cases and control subjects.

ELIGIBILITY:
Inclusion Criteria:

* new case of Behçet's disease available medical record Well known duration of BD, Well known current treatment used Well known current organ involvement

Exclusion Criteria:

* concomitant autoimmune or auto-inflammatory disorder; acute or chronic infections; cancer; diabetes; heart failure; gestation or up to six months after birth

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Sixty BD cases diagnosed by the International Study Group classification criteria for BD were included. BD cases were recruited from the outpatient clinic of Rheumatology and Rehabilitation Department, Mansoura University Hospitals. The study also included 60 age- and gender-matched normal subjects served as controls.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
BD activity was evaluated using BD Current Activity Form (BDCAF). | 3 years
  BD activity was assessed with BDCAF which assesse clinical characteristics present during the previous one month before evaluation. BDCAF include the following components: headaches; mouth ulcers; erythema; genital ulcers; arthritis; arthralgia; nausea/emesis/pain in abdomen; rectal bleeding; diarrhea; and new ocular, vascular, and nervous symptoms. Each component takes a score of (0) if absent or (1) if present [30]. The total BDCAF score was calculated by adding up the positive components (maximum score = 12). A BDCAF patient index score ≥2 was considered as active BD, while a score less than 2 was considered as inactive BD
Serum calprotectin concentrations | 3 years
  Blood samples were withdrawn from all participants 12 h after fasting. Samples underwent centrifugation at 4000 rpm for ten minutes. The sera were collected and kept at -80°C till analysis.
  Serum calprotectin concentrations were quantified utilizing a commercial calprotectin ELISA kit (Hycult Biotech Inc, US) based on manufacturer's instructions. Levels of high-sensitivity CRP (hsCRP) and albumin were detected using the immunoturbidimetric technique. Unit of measurment (μg/ml )
Ischaemia Modified Albumin (IMA) serum concentrations | 3 years
  IMA was quantified based on albumin cobalt binding colorimetric assay according to Bar-Or and colleagues and the levels were expressed in absorbance units (ABSU). To obtain corrected IMA values, the equation (individual albumin level/median albumin level of population) × IMA ABSU value was applied. Unit of measurment ( kU/L)

CONTACTS AND LOCATIONS:
Overall Officials: Sherin Mashaly, MD, Study Chair — Professor of Rheumatology and Rehabilitation
Locations (1):
- Mansoura University Hospital, Al Mansurah, Egypt